CLINICAL TRIAL: NCT00765414
Title: An Open-Label Extension Study of the Long-Term Safety and Efficacy of Recombinant Human Acid α-Glucosidase (rhGAA) Given as Enyzme Replacement Therapy to a Single Patient With Pompe Disease (Glycogen Storage Disease Type II) Who Were Previously Enrolled in Genzyme-Sponsored Enzyme Replacement Therapy Studies
Brief Title: Extension Study of Long-term Safety and Efficacy of Myozyme for a Single Patient With Pompe Disease Who Were Previously Enrolled in Genzyme Sponsored ERT Studies.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Medical Monitor, Genzyme Corporation
Organization: Sanofi (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AGLU02103
Record Dates: First submitted 2008-10-02; First posted 2008-10-03 (Estimated); Last update posted 2014-02-05 (Estimated); Status verified 2014-02

CONDITIONS: Pompe Disease Late-Onset; Glycogen Storage Disease Type II GSD II
MeSH Terms: interventions — GAA protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental)
  Interventions: Biological: Myozyme

INTERVENTIONS:
Biological: Myozyme — 30 mg/kg qow f and 40 mg/kg qow
  Other Names: Alglucosidase alfa

SUMMARY:
This extension study was to monitor the long-term safety and efficacy of rhGAA treatment in a single patient with infantile-onset Pompe disease who were previously treated with rhGAA in a Genzyme study.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent prior to participating in any study related procedures;
* Currently enrolled in Protocol AGLU01402
* Have the ability to comply with the clinical protocol, which required extensive clinical evaluations for an extended period of time.

Exclusion Criteria:

* Was pregnant or unwilling to use approved birth control during the course of the study;
* Had experienced any unmanageable AEs under Protocol AGLU01402 (as determined and agreed upon by the Principal Investigator and sponsor) due to rhGAA that would preclude continuing ERT;
* Was participating in any other investigational study.

Min Age: 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2003-04; Primary Completion 2006-04 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
The objective of this extension study was to monitor the long-term safety and efficacy of a single patient | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (1):
- University of Texas Health Science Center at San Antonio, San Antonio, Texas, United States